CLINICAL TRIAL: NCT05827237
Title: Primary Care Decision Rule for Chest Pain Using the Marburg Heart Score and Hs-troponin I Point of Care Test to Rule Out Acute Coronary Syndrome
Brief Title: Rule Out of ACS in Primary Care Using a Decision Rule for Chest Pain Including Hs-troponin I POCT
Acronym: POB HELP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Maastricht Universitair Medisch Centrum (Unknown); VieCuri Medical Centre (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Tobias N Bonten, MD PhD, Assistant professor, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: p20.013
Record Dates: First submitted 2023-03-21; First posted 2023-04-25 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Chest Pain; Myocardial Infarction; Acute Coronary Syndrome
Keywords: Chest pain; Primary care; General practice; Myocardial infarction; Troponin; Point of care test
MeSH Terms: conditions — Chest Pain; Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: A clustered randomized controlled trial in which general practices are randomized to the intervention- or control group in 2:1 ratio.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clinical decision rule (Experimental): Patients in whom the clinical decision rule is used to exclude acute coronary syndrome
  Interventions: Diagnostic Test: Clinical decision rule
- Standard care (No Intervention): Patients in whom the general practitioner decides upon referral following local guidelines.

INTERVENTIONS:
Diagnostic Test: Clinical decision rule — Clinical decision rule for acute chest pain, consisting of the Marburg Heart Score (5 questions) combined with a high-sensitive troponin I point of care test
  Arms: Clinical decision rule

SUMMARY:
The goal of this clustered, diagnostic randomized controlled trial is to study a clinical decision rule including a high-sensitive troponin I point of care test in patients with chest pain in primary care.

The main questions it aims to answer are:

1. Can unnecessary referrals to secondary care be reduced by the use of a clinical deci-sion rule in patients with new onset, non-traumatic chest pain in primary care? Compared to current daily practice.
2. What is the accuracy (sensitivity, negative prediction value) of the clinical decision rule for excluding ACS and MACE at 6 weeks and 6 months?

DETAILED DESCRIPTION:
This clustered, diagnostic randomized controlled trial will included patients with acute chest pain consulting their general practitioner. Practices in the intervention group will use a clinical decision rule consisting of the Marburg Heart Score and a high-sensitive troponin I point of care test to exclude acute coronary syndrome (ACS) and decide upon referral. Practices in the control group will apply usual care following local guidelines.

An independent endpoint committee consisting of a cardiologist and general practitioner will adjudicate the final diagnosis. Primary endpoints are ACS and Major Adverse Cardiac Events. A delayed reference standard of 6 months will be used.

For high sensitive troponin I measurement, the Siemens Atellica VTLi immunoassay analyser is used.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Acute chest pain
* Seen by general practitioner

Exclusion Criteria:

* <1 hour since onset of symptoms
* Inability to speak or understand Dutch
* Hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 946 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Hospital referral rate for acute chest pain | 24 hours after inclusion
  hospital referral rate for acute chest pain compared between intervention and control group
Hospital referral rate for acute chest pain | 6 weeks after inclusion
  hospital referral rate for acute chest pain compared between intervention and control group
Diagnostic accuracy of the clinical decision rule | 24 hours after inclusion
  Diagnostic accuracy (i.e. sensitivity, negative predictive value) for Acute Coronary Syndrome (ACS) and major adverse cardiac events (MACE).
  MACE is defined as a combined endpoint of ACS, percutaneous coronary intervention, coronary artery bypass grafting, coronary angiography revealing procedurally correctable stenosis managed conservatively and all-cause mortality.
Diagnostic accuracy of the clinical decision rule | 6 weeks after inclusion
  Diagnostic accuracy (i.e. sensitivity, negative predictive value) for ACS and major adverse cardiac events (MACE)
  MACE is defined as a combined endpoint of ACS, percutaneous coronary intervention, coronary artery bypass grafting, coronary angiography revealing procedurally correctable stenosis managed conservatively and all-cause mortality.
Diagnostic accuracy of the clinical decision rule | 6 months after inclusion
  Diagnostic accuracy (i.e. sensitivity, negative predictive value) for ACS and major adverse cardiac events (MACE)
  MACE is defined as a combined endpoint of ACS, percutaneous coronary intervention, coronary artery bypass grafting, coronary angiography revealing procedurally correctable stenosis managed conservatively and all-cause mortality.

SECONDARY OUTCOMES:
Cost-effectiveness | 6 months
  A trial-based cost analysis and a cost-utility analysis (costs per QALY, assessed using the EQ-5D-5L questionnaire)
Adherence to the recommendations of the clinical decision rule by general practitioners (GP) | 24 hours after inclusion
  Percentage of general practitioners following and deferring from the clinical decision rule, by comparing the GP's policy with the recommendations of the decision rule.
Patient reassurance measured by the State-Trait Anxiety Inventory | 1 week after inclusion
  Reassurance of patients, using the State-Trait Anxiety Inventory after the index consultation.
  State-Trait Anxiety Inventory: consisting of 40 self-report items on a 4-point Likert scale (min. 20- max. 80 points). Higher scores are correlated with higher levels of anxiety.
  Compared between intervention and control group.
Diagnostic accuracy of the gut feeling/ presence of a sense of alarm from general practitioners | 6 weeks after inclusion
  Diagnostic accuracy (i.e. sensitivity, negative predictive value) of general practitioner's gut feeling for Acute Coronary Syndrome and major adverse cardiac events (MACE). Using the Gut Feeling Questionnaire (GFC).
  The questionnaire consists of 11 items. The items use a 5-point Likert scale: completely disagree to completely agree. Items 1 and 11 are the same and ask the physician about their gut feeling: alarm vs reassuring.
  A high score indicates a sense of alarm
  (From Barais M, Fossard E, Dany A, et al. Accuracy of the general practitioner's sense of alarm when confronted with dyspnoea and/or chest pain: a prospective observational study. BMJ Open. 2020;10(2):e03434)
Diagnostic accuracy of the HEART-score | 6 weeks after inclusion
  Retrospectively for all patient with an ECG available for the occurrence of Acute Coronary Syndrome (ACS) and MACE.
  HEART-score assigning 0, 1 or 2 points to patient history, ECG abnormalities, Age, Cardiovascular risk factors and troponin. Lower score (0-3) indicates low risk for acute cardiac event.
  MACE is defined as a combined endpoint of ACS, percutaneous coronary intervention, coronary artery bypass grafting, coronary angiography revealing procedurally correctable stenosis managed conservatively and all-cause mortality.
Subgroup analyses for hospital referral rate for acute chest pain | 24 hours after inclusion
  Subgroups are classified by
  * sex
  * region (Leiden, Maastricht, Venlo)
  * socio-economic status (using postal-code)
  * duration of symptoms (<2 hours, 2-6 hours, 6-12 hours, >12 hours, >24 hours)
Subgroup analyses for hospital referral rate for acute chest pain | 6 weeks after inclusion
  Subgroups are classified by
  * sex
  * region (Leiden, Maastricht, Venlo)
  * socio-economic status (using postal-code)
  * duration of symptoms (<2 hours, 2-6 hours, 6-12 hours, >12 hours, >24 hours)
Subgroup analyses for diagnostic accuracy of the clinical decision rule | 24 hours after inclusion
  Subgroups are classified by
  * sex
  * region (Leiden, Maastricht, Venlo)
  * socio-economic status (using postal-code)
  * duration of symptoms (<2 hours, 2-6 hours, 6-12 hours, >12 hours, >24 hours)
  For the occurrence of ACS and MACE. MACE is defined as a combined endpoint of ACS, percutaneous coronary intervention, coronary artery bypass grafting, coronary angiography revealing procedurally correctable stenosis managed conservatively and all-cause mortality.
Subgroup analyses for diagnostic accuracy of the clinical decision rule | 6 weeks after inclusion
  Subgroups are classified by
  * sex
  * region (Leiden, Maastricht, Venlo)
  * socio-economic status (using postal-code)
  * duration of symptoms (<2 hours, 2-6 hours, 6-12 hours, >12 hours, >24 hours)
  For the occurrence of ACS and MACE. MACE is defined as a combined endpoint of ACS, percutaneous coronary intervention, coronary artery bypass grafting, coronary angiography revealing procedurally correctable stenosis managed conservatively and all-cause mortality.
Subgroup analyses for diagnostic accuracy of the clinical decision rule | 6 months after inclusion
  Subgroups are classified by
  * sex
  * region (Leiden, Maastricht, Venlo)
  * socio-economic status (using postal-code)
  * duration of symptoms (<2 hours, 2-6 hours, 6-12 hours, >12 hours, >24 hours)
  For the occurrence of ACS and MACE. MACE is defined as a combined endpoint of ACS, percutaneous coronary intervention, coronary artery bypass grafting, coronary angiography revealing procedurally correctable stenosis managed conservatively and all-cause mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Bonten, MD PhD, Principal Investigator — LUMC
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the main article, after deidentification (text, tables, figures and appendices)
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following main article publication
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] van den Bulk S, Petrus AHJ, Willemsen RTA, Boogers MJ, Meeder JG, Rahel BM, van den Akker-van Marle ME, Numans ME, Dinant GJ, Bonten TN. Ruling out acute coronary syndrome in primary care with a clinical decision rule and a capillary, high-sensitive troponin I point of care test: study protocol of a diagnostic RCT in the Netherlands (POB HELP). BMJ Open. 2023 Jun 8;13(6):e071822. doi: 10.1136/bmjopen-2023-071822. PMID 37290947
- See also: Up to date information about the study for patients and general practitioners (Dutch) — http://www.pobhelp.nl
- See also: Original registration on www.NTR.nl before start of the study — https://trialsearch.who.int/Trial2.aspx?TrialID=NL9525